CLINICAL TRIAL: NCT02463396
Title: Mindfulness Training Versus Treatment as Usual in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Mindfulness Training in Adults With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL48776.091.14; 837001501 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2015-05-19; First posted 2015-06-04 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2017-09

CONDITIONS: ADHD
Keywords: MBCT; Mindfulness; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (MBCT) for ADHD (Experimental): Adapted MBCT for ADHD
  Interventions: Behavioral: MBCT for ADHD
- Treatment as usual (TAU) (No Intervention): Usually medication & psycho-education

INTERVENTIONS:
Behavioral: MBCT for ADHD
  Arms: Mindfulness Based Cognitive Therapy (MBCT) for ADHD

SUMMARY:
The primary aim of this study is to investigate clinical effectiveness of mindfulness training versus treatment as usual (TAU) in adults with Attention Deficit Hyperactivity Disorder (ADHD). The secondary aim is to assess whether mindfulness training is cost-effective compared to TAU in adults with ADHD from a societal perspective.

DETAILED DESCRIPTION:
RATIONALE Attention Deficit Hyperactivity Disorder (ADHD) is a common neurodevelopmental disorder with a high persistence into adulthood. Patients with ADHD are primarily offered stimulant medication. However, not all patients are willing to take medication, some suffer from unacceptable side-effects and for many medication does not reduce their symptoms to the degree they would wish for. Therefore, there is a strong need for effective psychosocial interventions that are both accessible to a large group of patients and have been shown to be cost-effective, such as mindfulness training.

OBJECTIVE To examine the (cost)effectiveness of mindfulness versus treatment as usual (TAU) in adults with Attention Deficit Hyperactivity Disorder (ADHD).

HYPOTHESIS Mindfulness training will result in less ADHD symptoms, a better executive functioning, a better quality of life, and lower health care and societal costs.

STUDY DESIGN Randomised trial comparing mindfulness in addition to TAU with TAU alone. Baseline, end of treatment, follow-up 1 (6 months after baseline) and follow-up 2 (9 months after baseline) assessments will be done by blinded assessors and self-report questionnaires. After 9 months, patients allocated to the TAU condition will be offered mindfulness as well.

STUDY POPULATION N=120 adults with ADHD according to the DSM-5 using a structured psychiatric interview, referred to Radboudumc in Nijmegen, Reinier van Arkel in 's Hertogenbosch and Dimence in Deventer.

INTERVENTION The investigators have developed a treatment protocol of mindfulness for ADHD based on both the Mindfulness-Based Cognitive Therapy (MBCT) (Segal, Williams & Teasdale, 2013) and the mindfulness training for ADHD developed by Zylowska (2012).

STANDARD INTERVENTION TO BE COMPARED TO Treatment as usual, usually consisting of psychostimulants and psycho-education.

COST-EFFECTIVENESS ANALYSIS/ BUDGET IMPACT ANALYSIS Annual health care and societal cost savings are expected to be €1,2 million and €15,4 million, respectively.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include patients of 18 years and older who meet the following criteria:

* a primary diagnosis of ADHD, according to the criteria of Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV-TR) based on a structured Diagnostic Interview for ADHD, in adults (DIVA)
* capable of filling out questionnaires in Dutch

Exclusion Criteria:

* depressive disorder with psychotic symptoms or suicidality
* active manic episode
* borderline or antisocial personality disorder
* substance dependence
* autism spectrum disorder
* tic disorder with vocal tics
* learning difficulties or other cognitive impairments
* former participation in a MBCT or MBSR course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in investigator-rated ADHD symptoms | baseline, 3, 6 and 9 months
  Conners Adult ADHD Scale, investigator rating scale (CAARS-IR)

SECONDARY OUTCOMES:
Change from baseline in self-reported ADHD symptoms | baseline, 3, 6 and 9 months
  Conners Adult ADHD Scale, self-report version (CAARS-S)
Change from baseline in executive functioning | baseline, 3, 6 and 9 months
  Behavior Rating Inventory of Executive Function (BRIEF-A)
Change from baseline in patient functioning | baseline, 3, 6 and 9 months
  Outcome Questionnaire 45.2 (OQ 45.2)
Change from baseline in mindfulness skills | baseline, 3, 6 and 9 months
  Five Facet Mindfulness Questionnaire, short-form (FFMQ-SF)
Change from baseline in self-compassion | baseline, 3, 6 and 9 months
  Self-Compassion Scale, short-form (SCS-SF)
Change from baseline in positive mental health | baseline, 3, 6 and 9 months
  Mental Health Continuum, short-form (MHC-SF)
Change from baseline in health care consumption and productivity loss | baseline, 3, 6 and 9 months
  Trimbos/iMTA questionnaire for Costs associated with Psychiatric illness (TiC-P)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Janssen L, Kan CC, Carpentier PJ, Sizoo B, Hepark S, Schellekens MPJ, Donders ART, Buitelaar JK, Speckens AEM. Mindfulness-based cognitive therapy v. treatment as usual in adults with ADHD: a multicentre, single-blind, randomised controlled trial. Psychol Med. 2019 Jan;49(1):55-65. doi: 10.1017/S0033291718000429. Epub 2018 Feb 28. PMID 29486807
- [Derived] Janssen L, Kan CC, Carpentier PJ, Sizoo B, Hepark S, Grutters J, Donders R, Buitelaar JK, Speckens AE. Mindfulness based cognitive therapy versus treatment as usual in adults with attention deficit hyperactivity disorder (ADHD). BMC Psychiatry. 2015 Sep 15;15:216. doi: 10.1186/s12888-015-0591-x. PMID 26373634
- See also: Website Radboud University Medical Centre for Mindfulness — http://www.radboudcentrumvoormindfulness.nl/onderzoek/mindfulness-adhd/